CLINICAL TRIAL: NCT06979011
Title: Construction of Diagnostic Models for Pulmonary Hypertension Based on Novel Laboratory Indices and Echocardiogram Parameters
Brief Title: Construction of Clinical Diagnostic Model for Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2025-122-B; NSFC82270050 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; diagnosis; machine learning; heamodynamic status
MeSH Terms: conditions — Hypertension, Pulmonary; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pulmonary hypertension: people with pulmonary hypertension

SUMMARY:
Primary objective: To establish a non-invasive diagnostic model for pulmonary hypertension based on laboratory indicators and echocardiographic parameters.

Secondary objectives: To investigate the correlations between laboratory test indicators and echocardiographic data, and to develop new parameters based on preliminary analysis to assist in the diagnosis of pulmonary hypertension

DETAILED DESCRIPTION:
Data collection:

Collect vital signs (age, sex, etc.), clinical laboratory tests (complete blood count, biochemistry, BNP, D-dimer, and related derived parameters), and echocardiographic data from both the control group and pulmonary hypertension (PH) patients.

Obtain hemodynamic data measured via right heart catheterization (RHC) in PH patients.

Model development:

Construct a clinical diagnostic model using laboratory and echocardiographic data.

Fit hemodynamic parameters of PH patients based on their laboratory indicators, then assess the hemodynamic status using the fitted parameters and compare with actual measurements.

Secondary analyses:

Investigate correlations between echocardiographic parameters and laboratory test indicators in PH patients.

Identify core variables to develop novel diagnostic parameters and evaluate their diagnostic performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with any subtype of pulmonary hypertension (PH) confirmed by right heart catheterization (RHC) between 2020 and 2025.

No gender restrictions; age >18 years.

Availability of complete RHC records, transthoracic echocardiography (TTE), and laboratory test results (echocardiography and lab tests must be performed within one month before or after RHC).

Exclusion Criteria:

* Pulmonary veno-occlusive disease (PVOD)

Active or history of malignancy (or Malignant tumors if referring to current cases)

Hematologic disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with all types of PH
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
AUC | from 1 Jan 2025 to 30 Apr 2025
  the area under ROC curve

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No